CLINICAL TRIAL: NCT04587349
Title: Follow-up Study of the Effectiveness of Virtual Reality Therapy in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, 7400 Kaposvár, Tallián Gy. u 20-32, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB2020/06
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Stroke
Keywords: balance; movement; exergaming; posture; quality of life; gait
MeSH Terms: conditions — Stroke | interventions — Neurological Rehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise+FU 2/week (Active Comparator): Post stroke group that received 2 years of intensive therapy. (2/week)
  Interventions: Other: Neurorehabilitation
- Exercise+FU 3/week (Active Comparator): Post stroke group that received 2 years of intensive therapy. (3/week)
  Interventions: Other: Neurorehabilitation
- physiotherapy (Active Comparator): Post stroke group that received 2 years of traditional physiotherapy. (3/week)
  Interventions: Other: Physiotherapy
- Exercise+FU - controll (No Intervention): He did not receive treatment after 4 weeks of intensive care. it functions only as a control group.

INTERVENTIONS:
Other: Neurorehabilitation — Neurorehabilitation - 2 years-long intervention, targeted postural instability and mobility using at-limit intensity sensori and visuomotor agility training. (2/ week)
  Arms: Exercise+FU 2/week
Other: Neurorehabilitation — Neurorehabilitation - 2 years-long intervention, targeted postural instability and mobility using at-limit intensity sensori and visuomotor agility training. (3/ week)
  Arms: Exercise+FU 3/week
Other: Physiotherapy — Physiotherapy 2-years-long (3/week)
  Arms: physiotherapy

SUMMARY:
High intensity motion improves motor functions and quality of life in a neurologist. The investigators want to improve the clinical condition and quality of life of post-STROKE participants with a special sensory motor and visual motor agility therapy. High intensity motion improves engine function and quality of life in a neurologist. With special sensory motor and visual motility, investigaters want to improve the clinical condition and quality of life of STROKE participants. The investigaters randomly select participants who only perform the rehabilitation treatment have performed. The other group that will receive the study's control group will receive the traditional rehabilitation physiotherapy treatment. The investigaters assess the condition and quality of life of the patients. (EQ5-D, Barthel index, MRS test) The ivestigaters examine the functional movement and equilibrium variables of patients. (6MWT, Berg balance test, postgraduation) After that, participants are undergoing a 4-week intensive rehabilitation treatment. All participants are in post stroke. Primary Hypothesis will be changes in life-quality tests (EQ5-D, Barthel index, MRS test). Functional tests show progress 6MWT, Berg balance test and postural control testing with posturography. The results are compared and evaluated among the groups. The expected hypothesis is that visual and acoustic stimulation produces a better physical state at higher intensity. Patients were followed for 2 years and participated in a follow-up study every six months.

ELIGIBILITY:
Inclusion Criteria:

• post stroke

Exclusion Criteria:

* Sever heart problem
* sever demeanor
* alcoholism
* drug problems

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
gait / functional test | 2 years, m (higher point is better)
  6 minute walk test (m)
balance test | 2 years, (41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk )
  Berg Balance Test
postrural control test | 2 years, mm (2 year-long, the smaller the mm the better the result)
  posturography
Quality of life measured by EQ5-D scale | 2 years, 0-5 scale (2 year-long, higher point is better)
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. József Tollár, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=stroke+virtual+rehabilitation